CLINICAL TRIAL: NCT04153747
Title: High-power Short-duration Radiofrequency Application for Faster and Safer Pulmonary Vein Ablation Trial (POWER FAST III Trial)
Brief Title: High Radiofrequency Power for Faster and Safer Pulmonary Vein Ablation Trial (POWER FAST III)
Acronym: POWER-FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Dr. Sergio Castrejón-Castrejón, Electrophysiologist, Principal investigator (together with Dr. José Luis Merino), Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5064
Record Dates: First submitted 2019-11-02; First posted 2019-11-06 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Laser Speckle Contrast Imaging; Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional ablation (Active Comparator): Point-by-point catheter-based pulmonary veins isolation using convencional radiofrequency parameters.
  * Anterior aspect of pulmonary veins: 40 W, temperature limit 45 ºC, irrigation 17-30 ml/min; objective LSI>=6 or Ablation index >=500.
  * Posterior aspect of pulmonary veins: 20-40 W, temperature limit 45 ºC, irrigation 17-3 ml/min; objective LSI>=5 or Ablation index >=350.
  Interventions: Other: Low-power (25-40 W) radiofrequency ablation guided by lesion size index (LSI) and ablation index (AI) values; Other: Esophageal endoscopy; Diagnostic Test: Daily 30-seconds ECG
- High-power and short-duration ablation (Experimental): Point-by-point catheter-based pulmonary veins isolation using high-power and short duration radiofrequency: 70 W, duration per application 9-10 s (initial ramp 2-3 s according to the technical characterictics of radiofrequency sources), temperature limit 45 ºC, irrigation 17 ml/min, contac-force > 5 g.
  Interventions: Other: High-power and short-duration radiofrequency ablatio (70 W / 9-10 s); Other: Esophageal endoscopy; Diagnostic Test: Daily 30-seconds ECG

INTERVENTIONS:
Other: High-power and short-duration radiofrequency ablatio (70 W / 9-10 s) — Pulmonary veins electrical isolation: high-power and short-duration ablation
  Arms: High-power and short-duration ablation
Other: Low-power (25-40 W) radiofrequency ablation guided by lesion size index (LSI) and ablation index (AI) values — Pulmonary veins electrical isolation: low-power ablation.
  Arms: Conventional ablation
Other: Esophageal endoscopy — Esophageal endoscopy to detect postablation esophageal thermal lesions.
Diagnostic Test: Daily 30-seconds ECG — Transtelephonic daily 30-seconds single lead electrocardiogram
  Other Names: Transtelephonic daily 30-seconds single lead electrocardiogram

SUMMARY:
Multicenter 1:1 randomized study. Two atrial fibrillation ablation strategies are compared: 1) conventional ablation using point-by-point radiofrequency applications with power 40 W guided by LSI > 6 or AI > 500 on the anterior aspect of pulmonary veins and power 25 W guided by LSI >5 or AI >350 on the posterior wall near the esophagus; 2) point-by-point RF applications with power set at 70 W and duration 9-10 s. The main objective of the trial is the incidence of esophageal lesions evaluated with systematic endoscopy and clinical efficacy evaluated with daily ECG transtelephonic transmissions during 1-year follow-up. Secondary objectives include total RF time and parameters of acute PV isolation efficacy (first-pass isolation, acute reconnections and dormant conduction).

DETAILED DESCRIPTION:
Multicenter 1:1 randomized study: Hospital Universitario La Paz, Madrid; Hospital Clínico Universitario San Carlos, Madrid; Hospital Clínico y Provincial de Barcelona, Barcelona; Complejo Hospitalario de Navarra, Pamplona; Hospital Clínico Universitario de Valladolid; Hospital Clínico Universitario de Albacete; Hospital Clínico Universitario de Alicante; Hospital Universitario Virgen de las Nieves, Granada; Hospital La Fe, Valencia; Hospital Clínico de Valencia; Hospital Universitario Juan Ramón Jiménez, Huelva; Hospital de la Ribera, Alzira, Valencia. España. Spain.

Two atrial fibrillation ablation strategies are compared: 1) conventional ablation using point-by-point radiofrequency applications with power 40 W guided by LSI > 6 or AI > 500 on the anterior aspect of pulmonary veins and power 25-40 W guided by LSI >5 or AI >350 on the posterior wall near the esophagus; 2) point-by-point RF applications with power set at 70 W and duration 9-10 s.

The main objective of the trial is the incidence of esophageal lesions evaluated with systematic endoscopy and clinical efficacy evaluated with daily ECG transtelephonic transmissions during 1-year follow-up. Secondary objectives include total RF time and parameters of acute PV isolation efficacy (first-pass isolation, acute reconnections and dormant conduction).

Subestudy: asymptomatic cerebral lesions detected by 1,5 T MRI <72 h after ablation. Not all centers participate in the subestydy. However, if the center participates, all patients in both ablation groups will be included in the subestudy.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or persistent atrial fibrillation.
* Currently accepted class I or II indication for ablation according to practice guidelines: symptomatic arrhythmia, failure of at least 1 antiarrhythmic drug or patient's manifest preference of ablation instead of drugs.
* Age > 18 years.
* Acceptance of informed consent.

Exclusion Criteria:

* Previous pulmonary veins ablation of any type.
* Permanent atrial fibrillation or long-standing persistent AF (>1 year).
* Heart surgery <3 months before ablation.
* Coronary revascularization of any type <3 months before ablation.
* Myocardial infarction or acute coronary syndrome < 3 months before ablation.
* Stroke or transient cerebral ischaemic attack < 3 months before ablation.
* Persistent left atrial thrombus.
* Contraindication for anticoagulation.
* Absolute indication of double antiplatelet drugs.
* Complex congenital heart disease, corrected or not.
* Any clinical situation absolutely precluding an interventional procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Safety: incidence of esophageal thermal lesions | 24 hours after ablation (permissible up to 72 hours after ablation)
  Incidence of thermal esophageal lesions evaluated by endoscopy
Efficacy: recurrence of atrial arrhythmias | 1 year
  Recurrences of any atrial arrhythmias >30 seconds during 1-year follow-up evaluated by daily transtelephonic ECG transmissions (at least 1 ECG/day and additional transmissions whenever the patient perceives arrhythmia-related symptoms).
Total radiofrequency time | during ablation procedure
  Total radiofrequency time required for complete pulmonary veins isolation (included acute intraprocedural reconnections and dormant conduction).

CONTACTS AND LOCATIONS:
Overall Officials: José L Merino, PhD, Principal Investigator — Hospital Universitario La Paz, Madrid, España.; Sergio C Castrejón-Castrejón, PhD, Study Chair — Hospital Universitario La Paz, Madrid, España.; Carlos Escobar Cervantes, PhD, Study Chair — Hospital Universitario La Paz, Madrid, España.; Consuelo Froilán Torres, MD, Study Chair — Hospital Universitario La Paz, Madrid, España.; Andrés Fernández Prieto, MD, Study Chair — Hospital Universitario La Paz, Madrid, España.; Marcel Martínez Cossiani, MD, Study Chair — Hospital Universitario La Paz, Madrid, España.
Locations (1):
- University Hospital La Paz, Department of Cardiology, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castrejon-Castrejon S, Martinez Cossiani M, Basterra Sola N, Romero Roldan JD, Ibanez Criado JL, Osca J, Roca-Luque I, Moya A, Quesada A, Hidalgo Olivares VM, Perez Castellano N, Fernandez-Gomez JM, Macias-Ruiz R, Villanueva BB, Gonzalo Bada N, Froilan Torres C, Sanz Verdejo B, Sanchez Somonte P, Escobar Cervantes C, Moreno R, Merino JL; POWER FAST III Trial Investigators. High-Power Short-Duration Radiofrequency Application for Faster and Safer Pulmonary Vein Isolation: The POWER-FAST III Trial. JACC Clin Electrophysiol. 2025 Feb;11(2):350-361. doi: 10.1016/j.jacep.2024.10.009. Epub 2024 Dec 18. PMID 39708035